CLINICAL TRIAL: NCT02238392
Title: Arrhythmia Inducibility Versus Elimination of Dormant PV Conduction as a Procedural Endpoint of Catheter Ablation for Paroxysmal Atrial Fibrillation: a Prospective Randomized Trial
Brief Title: Adenosine vs AF Termination for Paroxysmal AF Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Rostock, Thomas Rostock, MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2014
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; pulmonary vein isolation; adenosine; AF terminatin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Adenosine testing after PVI and elimination of dormant conduction
  Interventions: Procedure: Adenosine test
- Group B - Termination of AF (Active Comparator): Termination of atrial fibrillation by catheter ablation
  Interventions: Procedure: Termination of AF

INTERVENTIONS:
Procedure: Adenosine test — Testing dormant conduction after PVI
  Arms: Group A
Procedure: Termination of AF — Testing AF iducibility and ermination of
  Arms: Group B - Termination of AF

SUMMARY:
This study investigates impact of adenosine versus AF inducibility and subsequent termination on the acute and long-term outcome of paroxysmal AF ablation.

DETAILED DESCRIPTION:
Despite intensive efforts to increase single procedure success rates of pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (AF), an arrhythmia-free surveillance has not raised beyond 80%. This prospective, randomized study investigates the efficacy of two different procedural endpoints in terms of single-procedure arrhythmia-free outcome.

A total number of 152 patients undergoing de-novo catheter ablation for paroxysmal AF will be randomized to two different treatment arms. In group-A patients, PVI will be performed with the patient either in spontaneous or induced AF. If AF will not terminate with PVI, ablation will be continued by targeting extra-PV AF sources with the desired endpoint of termination to sinus rhythm (SR). The ablation procedure in group-B patients consists of PVI exclusively, regardless to the underlying rhythm. In this group, all isolated PVs will be challenged to adenosine administration in the attempt to reveal and ablate dormant conduction. The primary endpoint is arrhythmia-free survival during a follow-up of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with paroxysmal AF
* de-novo AF ablation
* age > 18 years

Exclusion Criteria:

* persistent AF
* previous cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Arrhythmia-free survival | 1 year
  arrhythmia-free outcome during 1 year after the procedure

SECONDARY OUTCOMES:
Recurrence if PV conduction after ablation in PVs with abolished dormant conduction | 1 year
  PV conduction recurrences after elimination of dormant conduction. This endpoint will be evaluated during repeat procedures for recurrences of atrial fibrillation or atrial tachycardia.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rostock, MD, Principal Investigator — University Hospital Mainz, Dept. of Cardiology
Locations (1):
- University Hospital Mainz, Department of Medicine II, Mainz, Germany

REFERENCES:
- [Derived] Theis C, Konrad T, Mollnau H, Sonnenschein S, Kampfner D, Potstawa M, Ocete BQ, Bock K, Himmrich E, Munzel T, Rostock T. Arrhythmia Termination Versus Elimination of Dormant Pulmonary Vein Conduction as a Procedural End Point of Catheter Ablation for Paroxysmal Atrial Fibrillation: A Prospective Randomized Trial. Circ Arrhythm Electrophysiol. 2015 Oct;8(5):1080-7. doi: 10.1161/CIRCEP.115.002786. Epub 2015 Aug 21. PMID 26297786